CLINICAL TRIAL: NCT05926739
Title: Prospective Evaluation of the Performance and Safety of the PHENIX LIBERTY, a Medical Device for Electrostimulation and Biofeedback, in the Treatment of Locomotor Disorders
Brief Title: Performance and Safety of the PHENIX LIBERTY, a Medical Device for Electrostimulation and Biofeedback, in the Treatment of Musculoskeletal Disorders
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vivaltis (Industry)
Collaborators: CEISO (Industry); Human Physio (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2023-A02460-45
Record Dates: First submitted 2023-06-22; First posted 2023-07-03 (Actual); Last update posted 2024-12-24 (Actual); Status verified 2024-12

CONDITIONS: Musculoskeletal Disorder
Keywords: Electrical stimulation; Biofeedback; Knee; Low Back Pain
MeSH Terms: conditions — Musculoskeletal Diseases; Low Back Pain | interventions — Electric Stimulation; Biofeedback, Psychology

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Standard of care plus additional questionaire (Other): As part of this clinical investigation, the medical device under investigation is used in accordance with its usual use, and the patient's therapeutic procedure includes additional, non-invasive procedures. These additional procedures relate to the addition of an endof- life visit and validated questionnaires assessing functional deficiencies and impact on daily life.
  Interventions: Device: Electrical stimulation and biofeedback with Phenix Liberty medical device

INTERVENTIONS:
Device: Electrical stimulation and biofeedback with Phenix Liberty medical device — 12 sessions of electrical stimulation and biofeedback performed between 6 and 8 weeks at regular intervals according to a schedule drawn up by the physiotherapist.
  The patient will undergo 12 therapeutic functional reeducation sessions, at regular intervals according to a schedule drawn up by the physiotherapist, during which the PHENIX LIBERTY device may be used. The patients will complete questionnaires at the end of the care.
  Overall, the functional rehabilitation sessions will include muscle testing, electrostimulation and biofeedback.
  The follow up will be conduct as follow :
  * 12 sessions between 6 and 8 weeks
  * 1 end visit, within the week after the 12th session

SUMMARY:
Evaluate the evolution of locomotor abilities in patients treated with functional electrostimulation and biofeedback (PHENIX LIBERTY VIVALTIS device) for musculoskeletal disorders of the knee and spine.

Does the use of the medical device in the treatment of musculoskeletal disorders lead to an improvement ?

Participants will use the medical device, which provides electrical stimulation, biofeedback and pressure biofeedback to re-educate the muscles of the knee and spine area and

DETAILED DESCRIPTION:
Rational :

Today, musculoskeletal disorders (MSDs) are considered to be one of the world's leading pathologies. They are also the most widespread occupational pathology in Europe. MSDs include a variety of conditions affecting bones, joints, muscles and connective tissues. To treat these disorders, the guidelines recommend non-drug therapies as first-line treatments for chronic low-back pain and osteoarthritis pain, such as electrostimulation and biofeedback therapy.

In this context, the promoter wishes to carry out this study in order to reinforce the data currently available on the medical device PHENIX LIBERTY.

Design:

Prospective, interventional with non invasive and non burdensome procedure, non-comparative, multicenter, open-label study of a CE-marked medical device

Intervention :

As part of this clinical investigation, the medical device under investigation is used in accordance with its usual use, and the patient's therapeutic procedure includes additional, non-invasive procedures. These additional procedures relate to the addition of an end-of-life visit and validated questionnaires assessing functional deficiencies and impact on daily life.

The care will be conduct as follow:

* 1 inclusion visit (V0) (from 1 say to 15 days prior the the first functionnal therapeutic re-education session)
* 12 sessions of functional therapeutic re-education, during which the PHENIX LIBERTY device may be used. Sessions performed at regular intervals according to a schedule drawn up by the physiotherapist (between 6 and 8 weeks);
* 1 end visit (V13), 1 week after the 12th session to complet questionnaires

In total, the patient will be followed 11 weeks maximum

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (between 18 and 65 years of age);
* Patient presenting at least one of the following symptoms related to a locomotor disorder of the knee and/or spine: pain, hypertonia, amyotrophy, mobility restriction, muscle weakness, reduction or loss of motor control, reduction in motor pattern, trophic anomaly;
* Patient able to make himself available to attend sessions regularly and is confident of being able to complete all sessions; ;
* Patient who has signed the study participation consent form;y;
* Patient physically and mentally willing and able, according to the investigator's judgment at the time of recruitment, to perform the procedures under study;
* Patient with social security coverage.

Exclusion Criteria:

* Patients with Stroke, Alzheimer's, multiple sclerosis, peripheral nervous system disorders, spinal cord injury or with cognitive and/or behavioural disorders likely, in the practitioner's judgement in the practitioner's judgement, interact with the self-assessment or biofeedback;
* Patients with hypersensitivity to electrostimulation;
* Patients who, in the 1 month prior to inclusion, have had injections of corticosteroids (e.g. hyaluronate) in the knee/spine concerned;
* Patients with an implanted pacemaker or spinal cord pacemaker;
* Pregnant at the time of the inclusion visit, or wishing to become pregnant during the treatment period;
* Patients who have renounced their liberty by administrative or judicial sentence, or under guardianship or limited judicial protection;
* Patient participating in another interventional clinical trial for the same pathology or testing/having tested an investigational drug in the 30 days prior to inclusion in the study;
* Patient unable to read or write French;

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2024-08-19 (Actual); Primary Completion 2024-12-18 (Actual); Study Completion 2024-12-18 (Actual)

PRIMARY OUTCOMES:
Mean change in Lower Extremity Functional Scale (LEFS) score on the impact of locomotor disorders of the knee | At Day 0 and Week 11 (at the end visit within the week after the 12th seance)
  The Lower Extremity Functional Scale (LEFS) is used by physiotherapists and occupational therapists in many clinical settings. It is an English-language measurement tool that collects psychometric data and assesses the functional status of the lower limbs. It consists of 20 questions on the level of difficulty experienced during everyday activities.
Mean change in the Oswestry Disability Index (ODI) score for the impact of locomotor disorders of the spine. | At Day 0 and Week 11 (at the end visit within the week after the 12th seance)
  The ODI will be used to assess the disability caused by Lower Back Pain (LBP)
  The Oswestry Disability Index (ODI), a patient-completed questionnaire that gives a subjective percentage score of the level of function (disability) in activities of daily living in people undergoing rehabilitation after low back pain. The questionnaire examines the level of disability in 10 activities of daily living. Each item consists of 6 statements rated from 0 to 5. With 0 indicating the lowest level of disability and 5 the highest, the total score is calculated as a percentage, with 0% indicating no disability and 100% indicating the highest level of disability.

SECONDARY OUTCOMES:
Change in patients' visual analog scale (VAS) pain scores for knee pain and/or spine pain at rest and on palpation | At Day 0 and Week 11 (at the end visit within the week after the 12th seance)
  The pain caused by the TMS of the knee and/or the spine will be assessed by the Visual Analogue Scale (VAS).
  The VAS is made up of a 10-centimeter line anchored by two ends of the pain. 10 is the first end being the "maximum pain imaginable" and 0 is the other end being "no pain"
Trends in consumption of painkillers and anti-inflammatories | At Day 0 and Week 11 (at the end visit within the week after the 12th seance)
  Rate of consuption of painkillers and anti-inflammatories
Changes in the rate of improvement of hypertonia of the concerned area (knee or spine) through measurement of myoelectric activity | At Day 0 and Week 11 (at the end visit within the week after the 12th seance)
  A surface Electromyography (EMG) will be used. Muscle electrical activity provides a "map" of muscle recruitment according to exercise conditions (position, relative load, type of resistance, type of support, etc.).
Changes in the rate of improvement of hypertonia of the concerned area (knee or spine) through Oxford Grading Scale | At Day 0 and Week 11 (at the end visit within the week after the 12th seance)
  The Oxford scale is commonly used to manually assess muscle strength, and can help diagnose problems in which weakness plays a role. According to the Oxford scale, muscle strength is rated from 0 to 5 (0 being no muscle contraction > 5 being movement through a full range against full resistance). Scoring is as follows: 0 → No visible or palpable contraction, 1 → Visible/palpable muscle contraction but no movement, 2 → Movement across full range with gravity eliminated (low strength), 3 → Movement across full range against gravity only (fair strength), 4 → Movement across full range against gravity with some resistance (good strength), 5 → Movement across full range against gravity with full resistance (normal strength).
Changes in the rate of improvement in awakening and muscle strengthening through Oxford grading scale | At Day 0 and Week 11 (at the end visit within the week after the 12th seance)
  The Oxford scale is commonly used to manually assess muscle strength, and can help diagnose problems in which weakness plays a role. According to the Oxford scale, muscle strength is rated from 0 to 5 (0 being no muscle contraction > 5 being movement through a full range against full resistance). Scoring is as follows: 0 → No visible or palpable contraction, 1 → Visible/palpable muscle contraction but no movement, 2 → Movement across full range with gravity eliminated (low strength), 3 → Movement across full range against gravity only (fair strength), 4 → Movement across full range against gravity with some resistance (good strength), 5 → Movement across full range against gravity with full resistance (normal strength).
Changes in the rate of improvement in awakening and muscle strengthening through measurement of myoelectric activity | At Day 0 and Week 11 (at the end visit within the week after the 12th seance)
  A surface Electromyography (EMG) will be used. Muscle electrical activity provides a "map" of muscle recruitment according to exercise conditions (position, relative load, type of resistance, type of support, etc.).
Changes of microcirculation of the concerned spine area | At Day 0 and Week 11 (at the end visit within the week after the 12th seance)
  Assessment on the basis of clinical palpation examination done by the practitioner
Changes of the microcirculation of the concerned knee area | At Day 0 and Week 11 (at the end visit within the week after the 12th seance)
  The measurement of the muscular perimeter around the concerned knee will be assessed by a tape measure
Changes of the improvement of the motor control through the measurement of myoelectrical activity | At Day 0 and Week 11 (at the end visit within the week after the 12th seance)
  A surface Electromyography (EMG) will be used. Muscle electrical activity provides a "map" of muscle recruitment according to exercise conditions (position, relative load, type of resistance, type of support, etc.).
Change in patient's quality of life | At Day 0 and Week 11 (at the end visit within the week after the 12th seance)
  The SF-36 will be used to assess the quality of life score.
  The SF-36, as described in the name, is a 36-item patient-reported questionnaire that covers eight health domains: physical functioning (10 items), bodily pain (2 items), role limitations due to physical health problems (4 items), role limitations due to personal or emotional problems (4 items), emotional well-being (5 items), social functioning (2 items), energy/fatigue (4 items), and general health perceptions (5 items). Scores for each domain range from 0 to 100, with a higher score defining a more favorable health state.
Pecentage of patients with an improvement in locomotor disorders | At Day 0 and Week 11 (at the end visit within the week after the 12th seance)
  This outcome will be assessed according to the practitioner's opinion. Does the practitioner think that an improvement has been observed --> Yes / No ?
Incidence of adverse events | At Day 0 and Week 11 (at the end visit within the week after the 12th seance)
  Rate of the incidence of adverse events related to the medical device
Evaluation of responses to the patient satisfaction questionnaire on the use of the PHENIX LIBERTY device after therapeutic management | At Day 0 and Week 11 (at the end visit within the week after the 12th seance)
  The satisfaction questionnaire is constructed on the basis of the Likert Scale. The sponsor has written an questionnaire regarding the use of the Phenix Liberty for the patient. The Likert scale (or attitude scale) is a semantic rating system, generally consisting of 5 or 7 items, used in surveys to measure and evaluate perceptions, attitudes and opinions. The evaluation will be based on the following responses: Strongly agree (=5) ; Agree (=4) ; Rather agree (=3) ; Rather disagree (=2) ; Disagree (=1= ; Strongly disagree (=0). The minimum score 0 means a worse outcome and the maximum score 5 means a better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Mathias Willame, Principal Investigator — Human Physio
Locations (1):
- Human Physio, Nîmes, France